CLINICAL TRIAL: NCT04982315
Title: Pragmatic Trial of Acupuncture for Chronic Low Back Pain in Older Adults
Brief Title: Acupuncture for Chronic Low Back Pain in Older Adults
Acronym: BackInAction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BackInAction; UH3AT010739 (NIH)
Record Dates: First submitted 2021-07-01; First posted 2021-07-29 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low-back Pain; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Acupuncture (Experimental): Participants randomized to standard acupuncture will receive 8-15 acupuncture treatments over 3 months.
  Interventions: Procedure: Standard Acupuncture
- Enhanced Acupuncture (Experimental): Participants randomized to enhanced acupuncture will receive 12-21 acupuncture treatments over 6 months.
  Interventions: Procedure: Enhanced Acupuncture
- Usual Care (No Intervention): Participants assigned to the usual care arm will not receive acupuncture and will be asked to not get acupuncture over the one-year course of the study.

INTERVENTIONS:
Procedure: Standard Acupuncture — The standard acupuncture intervention is based on classical Chinese acupuncture therapy. Participants randomized to standard acupuncture will receive up to 15 acupuncture treatments over 3 months with the total number being determined by the patient and acupuncturist together. All treatments will include acupuncture needling only. They will be provided at medical facilities or in private acupuncturists' offices.
  Arms: Standard Acupuncture
Procedure: Enhanced Acupuncture — The enhanced acupuncture intervention includes the 3 months of standard acupuncture plus an additional 3 months of maintenance acupuncture. Participants randomized to enhanced acupuncture will receive up to 21 acupuncture treatments over 6 months. The maintenance acupuncture treatment sessions are expected to consist of the same intervention used in the first 3 months of care described in the standard acupuncture arm, plus up to 6 treatments during the maintenance phase. All treatments will include acupuncture needling only. They will be provided at medical facilities or in private acupuncturists' offices.
  Arms: Enhanced Acupuncture

SUMMARY:
The main goal of the BackInAction research study is to determine the effectiveness of a standard course of acupuncture (15 sessions of acupuncture over 3 months) and an enhanced course of acupuncture (an additional 6 sessions of acupuncture over months 4-6) in improving back-related disability in older adults (65+ years) with chronic low back pain compared to usual care alone. Key secondary aims are to determine the effectiveness of acupuncture in improving a composite score of pain intensity and pain interference.

DETAILED DESCRIPTION:
Background: A critical gap exists in evidence regarding the safety and effectiveness of treatments for older adults (65+ years) with chronic low back pain. Acupuncture has been found to be effective in treating chronic low back pain in younger adults. Yet trials have rarely included older adults, who have more comorbidities and may respond differently than typical trial participants. BackInAction has been designed to address this gap.

Purpose: The main goal of BackInAction is to evaluate the effectiveness of a standard course of acupuncture (up to 15 sessions of acupuncture over 3 months) and an enhanced course of acupuncture (up to an additional 6 sessions of acupuncture over months 4-6) in improving back-related disability in older adults with chronic low back pain compared to usual care alone. Key secondary aims are to determine the effectiveness of acupuncture in improving a composite score of pain intensity and pain interference.

Design and Outcomes: In this pragmatic, three-arm parallel groups multi-site randomized controlled trial, the investigators will recruit and randomize at least 789 adults ≥ 65 years of age with chronic low back to standard acupuncture, enhanced acupuncture, or usual medical care alone in four health-care systems. These include two integrated health care systems, a fee-for-service system and a network of federally qualified health centers. Primary outcome data will be collected by questionnaire at 3-, 6-, and 12-months post-randomization. In addition, short monthly surveys will capture data on physical function and a composite score of pain intensity and pain interference.

Interventions and Duration: Standard acupuncture will consist of 3 months (90 days) of acupuncture needling, with a proposed minimum of 8 treatments and a maximum of 15. Enhanced acupuncture will include the standard acupuncture plus an additional 3-month maintenance period, with a maximum of six additional treatments. Usual medical care will consist of the care that individuals receive according to their insurance benefits plus anything else they pay for out of pocket. The investigators will ask those assigned to usual medical care to avoid acupuncture for the year they are enrolled in the study. Both active treatment arms will also have access to usual medical care. Participants will be enrolled in the study for 12 months.

Sample Size and Population: BackInAction will include patients at least 65 years of age with uncomplicated chronic low back pain with or without radiculopathy. The investigators plan to enroll at least 789 participants (263 per study arm). Participants will be recruited from four health plans, with varying numbers of participants from each site. Randomization will be stratified by health care system, age category and gender. The investigators expect the racial and ethnic mix will roughly parallel that of the older Medicare population.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 65 years of age
* Is a current member or patient of the healthcare system
* Visited a health care provider for low back pain within the past 12 months
* Received primary care at one of the participating health care systems
* Has back pain that is uncomplicated with or without radicular pain
* Back pain at least 3 months
* General activity question from PEG (Pain, Pain Interference with Enjoyment, General Activity scale) at least 3
* Primary care provider provides permission to contact patient
* Willing and able to provide consent (Callahan cognitive impairment screener at least 3)

Exclusion Criteria:

* Specific types of back pain (metastatic cancer or bone cancer or secondary cancers, vertebral fractures, spinal infection, active inflammatory disease)
* Low back surgery within past 3 months
* Receiving workers compensation or involved in litigation related to chronic low back pain
* Acupuncture within the last 6 months
* Does not speak or write English or Spanish
* Major psychosis, dementia
* Current cancer treatment
* Red flags of serious underlying illness (a fever most days in the last month; recent unexplained weight loss of 10 lbs or more)
* Living in a nursing home, on Hospice, or palliative care
* Non-speaking deafness
* Non-reliable transportation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 807 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn L DeBar, PhD, MPH, Principal Investigator — Kaiser Permanente; Andrea J Cook, PhD, Principal Investigator — Kaiser Permanente
Locations (4):
- United States (4):
  - Kaiser Permanente Division of Research, Oakland, California
  - Sutter Health, Walnut Creek, California
  - Institute for Family Health, New York, New York
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Kaiser Permanente Washington-based data coordinating center will produce a releasable de-identified database corresponding to the primary outcomes manuscript that can be used by research investigators outside of the study. This dataset will also include the NIH HEAL (Helping to End Addiction Long-term) Initiative common data elements collected from study participants. The dataset will be completely de-identified in accordance with the definitions provided in the Health Insurance Portability and Accountability Act and in accordance to the standards set forth in the Department of Health and Human Services Regulations for the Protection of Human Subjects. All identifiers specified in HIPAA will be recoded in a manner that will make it impossible to deduce or impute the specific identity of any patient. The database will not contain any institutional or healthcare system identifiers.
Supporting Information: Study Protocol
Time Frame: The de-identified dataset will be released within 12 months of the publication of the primary manuscript.
Access Criteria: Access to the de-identified database housed in an NIH-assigned repository will be in accordance with procedures and regulations of the NIH HEAL Initiative and the project funder (NCCIH). The project team does not plan to provide any support for investigators using the HEAL releasable database.
URL: https://heal.nih.gov/about/public-access-data

REFERENCES:
- [Derived] DeBar LL, Wellman RD, Justice M, Avins AL, Beyrouty M, Eng CM, Herman PM, Nielsen A, Pressman A, Stone KL, Teets RY, Cook AJ. Acupuncture for Chronic Low Back Pain in Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2531348. doi: 10.1001/jamanetworkopen.2025.31348. PMID 40938602
- [Derived] Justice M, Piccorelli A, Avins AL, Cook AJ, Eng CM, Nielsen A, Pressman A, Stone KL, Teets RY, Wellman R, DeBar LL. Baseline sample characteristics for the BackInAction pragmatic trial of acupuncture for chronic low back pain in older adults. Contemp Clin Trials. 2025 Aug;155:107981. doi: 10.1016/j.cct.2025.107981. Epub 2025 Jun 6. PMID 40484274
- [Derived] Wang PZ, Pressman A, Sanchez G, Aparicio C, Nielsen A, Avins A. Prior acupuncture experience among elderly participants enrolled in a clinical trial of acupuncture for chronic low back pain: Implications for future trials. Integr Med Res. 2024 Jun;13(2):101042. doi: 10.1016/j.imr.2024.101042. Epub 2024 Apr 17. PMID 38765784
- [Derived] DeBar LL, Justice M, Avins AL, Cook A, Eng CM, Herman PM, Hsu C, Nielsen A, Pressman A, Stone KL, Teets RY, Wellman R. Acupuncture for chronic low back pain in older adults: Design and protocol for the BackInAction pragmatic clinical trial. Contemp Clin Trials. 2023 May;128:107166. doi: 10.1016/j.cct.2023.107166. Epub 2023 Mar 27. PMID 36990274

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic low back pain that had persisted for >3 months were recruited from four different health systems. The first participant was enrolled in August 2021 and the last participant was enrolled October 2022.
Pre-assignment Details: Of 12,438 participants screened for eligibility, 800 were randomized and enrolled in the study.
Period: Overall Study
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Started | 266 | 265 | 269
3-Month Survey | 218 | 247 | 252
6-Month Survey | 223 | 247 | 248
12-Month Survey | 220 | 244 | 239
Completed | 237 | 260 | 256
Not Completed | 29 | 5 | 13
Not completed — Death | 1 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Withdrawal by Subject | 24 | 1 | 2
Not completed — Dealing with health/life issues | 3 | 4 | 7
Not completed — Privacy concerns | 1 | 0 | 0
Not completed — Withdrawal by research team | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants with chronic low back pain that had persisted for >3 months were recruited from four different health systems. The first participant was enrolled in August 2021 and the last participant was enrolled October 2022.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture | Total
Number analyzed (Participants) | 266 | 265 | 269 | 800
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 266 | 265 | 269 | 800
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.7 (6.0) | 73.4 (5.8) | 73.8 (6.1) | 73.6 (6.0)
Age, Customized [Count of Participants; unit: Participants]
  65-74 years old | 157 | 159 | 156 | 472
  75-84 years old | 94 | 95 | 98 | 287
  85+ years old | 15 | 11 | 15 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 164 | 164 | 495
  Male | 99 | 101 | 105 | 305
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 33 | 28 | 85
  Not Hispanic or Latino | 230 | 217 | 227 | 674
  Unknown or Not Reported | 12 | 15 | 14 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 1 | 6
  Asian | 14 | 16 | 13 | 43
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 0 | 3
  Black or African American | 41 | 55 | 43 | 139
  White | 187 | 159 | 186 | 532
  More than one race | 4 | 9 | 5 | 18
  Unknown or Not Reported | 14 | 24 | 21 | 59
Education [Count of Participants; unit: Participants] — Formal education background Population: Missing data for 2 participants
  Participants
    HS Diploma or less: number analyzed (Participants) | 266 | 264 | 268 | 798
    HS Diploma or less | 33 | 36 | 38 | 107
    At least some college: number analyzed (Participants) | 266 | 264 | 268 | 798
    At least some college | 147 | 154 | 141 | 442
    College graduate or higher degree: number analyzed (Participants) | 266 | 264 | 268 | 798
    College graduate or higher degree | 86 | 74 | 89 | 249
Clinical Site [Count of Participants; unit: Participants] — Research project clinical site.
  Participants
    IFH | 39 | 42 | 42 | 123
    KPNC | 96 | 93 | 97 | 286
    KPWA | 62 | 62 | 61 | 185
    Sutter | 69 | 68 | 69 | 206
Household Income [Count of Participants; unit: Participants] — Population: Missing data for 38 participants.
  Participants
    Less than $25,000: number analyzed (Participants) | 261 | 260 | 241 | 762
    Less than $25,000 | 30 | 37 | 32 | 99
    $25,000 - $49,999: number analyzed (Participants) | 261 | 260 | 241 | 762
    $25,000 - $49,999 | 47 | 42 | 35 | 124
    $50,000 - $99,999: number analyzed (Participants) | 261 | 260 | 241 | 762
    $50,000 - $99,999 | 77 | 79 | 67 | 223
    $100,000 - $149,999: number analyzed (Participants) | 261 | 260 | 241 | 762
    $100,000 - $149,999 | 64 | 72 | 76 | 212
    $150,000 or more: number analyzed (Participants) | 261 | 260 | 241 | 762
    $150,000 or more | 43 | 30 | 31 | 104
Received Disability for Lower Back Pain [Count of Participants; unit: Participants] | 29 | 24 | 24 | 77
Married or Domestic Partnered [Count of Participants; unit: Participants] | 156 | 147 | 152 | 455
Pain Limits Work [Count of Participants; unit: Participants] — Population: Missing data for 2 participants
  Participants
    Never: number analyzed (Participants) | 265 | 265 | 268 | 798
    Never | 13 | 12 | 8 | 33
    Some Days: number analyzed (Participants) | 265 | 265 | 268 | 798
    Some Days | 134 | 122 | 120 | 376
    Most Days: number analyzed (Participants) | 265 | 265 | 268 | 798
    Most Days | 71 | 79 | 78 | 228
    Every Day: number analyzed (Participants) | 265 | 265 | 268 | 798
    Every Day | 47 | 52 | 62 | 161
BMI [Count of Participants; unit: Participants] — Population: Missing data for 12 participants
  Participants
    Underweight (<18.5 kg.m2): number analyzed (Participants) | 261 | 263 | 264 | 788
    Underweight (<18.5 kg.m2) | 3 | 4 | 4 | 11
    Normal (18.5 - <25 kg/m2): number analyzed (Participants) | 261 | 263 | 264 | 788
    Normal (18.5 - <25 kg/m2) | 73 | 80 | 85 | 238
    Overweight (25 - <30 kg/m2): number analyzed (Participants) | 261 | 263 | 264 | 788
    Overweight (25 - <30 kg/m2) | 99 | 94 | 93 | 286
    Obese (>=30 kg/m2): number analyzed (Participants) | 261 | 263 | 264 | 788
    Obese (>=30 kg/m2) | 86 | 85 | 82 | 253
BMI Mean [Mean (Standard Deviation); unit: kg/m^2] — Population: Missing BMI data for 12 participants
  kg/m^2
    number analyzed (Participants) | 261 | 263 | 264 | 788
    (all) | 28.4 (6.4) | 28.1 (6.0) | 28.0 (5.9) | 28.1 (6.1)
Frailty [Count of Participants; unit: Participants] — The frailty scale used a modified version of the 5-item questionnaire by Morley, et al. Participants were asked four yes-no questions pertaining to fatigue, difficulty climbing stairs, difficulty walking and weight loss of more than 5% in the last year. The fifth item used EHR data to indicate the present of five of eleven predefined illnesses. Each item was coded as 1 for yes and 0 for no. The frailty score was calculated as the sum of the five items, yielding a range of 0 (best) to 5 (worst). Frailty scores correspond to the following categories: 0=Robust health, 1-2=Pre-frail, 3-5=Frail. Population: Missing complete data for 33 participants
  Participants
    Robust Health: number analyzed (Participants) | 257 | 255 | 255 | 767
    Robust Health | 82 | 63 | 78 | 223
    Pre-Frailty: number analyzed (Participants) | 257 | 255 | 255 | 767
    Pre-Frailty | 126 | 134 | 128 | 388
    Frailty: number analyzed (Participants) | 257 | 255 | 255 | 767
    Frailty | 49 | 58 | 49 | 156
Frailty Mean [Mean (Standard Deviation); unit: units on a scale] — Mean of Frailty (description above). The frailty score was calculated as the sum of the five items, yielding a range of 0 (best) to 5 (worst). Frailty scores correspond to the following categories: 0=Robust health, 1-2=Pre-frail, 3-5=Frail. Population: Missing data for 33 participants.
  units on a scale
    number analyzed (Participants) | 257 | 255 | 255 | 767
    (all) | 1.3 (1.2) | 1.5 (1.2) | 1.3 (1.2) | 1.4 (1.2)
Medical Morbidity (Elixhauser) [Mean (Standard Deviation); unit: units on a scale] — Scale range from 0-13; a higher score always indicates a greater comorbidity burden. Population: Missing data for 2 participants
  units on a scale
    number analyzed (Participants) | 265 | 264 | 269 | 798
    (all) | 2.4 (1.9) | 2.6 (2.1) | 2.5 (2.1) | 2.5 (2.0)
Any Opioid in Prior 3 Months [Count of Participants; unit: Participants] | 44 | 35 | 31 | 110
Long-term Opioid Therapy [Count of Participants; unit: Participants] — Long-term opioid therapy (60-day supply in the last 3 months)
  Participants | 14 | 7 | 3 | 24
Multiple Musculoskeletal Pain Conditions [Count of Participants; unit: Participants] — Musculoskeletal conditions include following ICD diagnostic codes within last year: back pain; neck pain; fibromyalgia; limb/extremity, joint, and non-systematic noninflammatory pain; muculoskeletal chest pain, headache, jaw pain, and general pain. (from the EHR)
  Participants | 224 | 220 | 243 | 687
Number of Musculoskeletal Pain Conditions [Mean (Standard Deviation); unit: Number of conditions] — Number of Musculoskeletal Pain Conditions (from the EHR)
  Number of conditions | 1.6 (1.1) | 1.7 (1.2) | 1.7 (1.0) | 1.7 (1.1)
Types of Painful Conditions [Count of Participants; unit: Participants] — Types of Painful Conditions (from the EHR)
  Participants
    Back pain | 229 | 228 | 250 | 707
    Neck pain | 59 | 60 | 43 | 162
    Fibromyalgia | 2 | 6 | 5 | 13
    Limb/extremity, joint, and non-systemic, non-inflammatory arthritic pain | 175 | 176 | 197 | 548
    Musculoskeletal chest pain | 36 | 38 | 34 | 108
    Headache or migraine | 26 | 19 | 22 | 67
    Toothache, ear or jaw pain | 3 | 8 | 6 | 17
    General pain | 127 | 134 | 147 | 408
Substance Use Disorder Diagnosis [Count of Participants; unit: Participants] — Substance Use Disorder Diagnosis (from the EHR)
  Participants
    Substance use disorder | 6 | 8 | 4 | 18
    Opioid use disorder | 2 | 1 | 1 | 4
    Stimulant use disorder | 0 | 0 | 1 | 1
    Sedative use disorder | 0 | 0 | 2 | 2
    Alcohol use disorder | 3 | 8 | 0 | 11
    Cannabis use disorder | 2 | 1 | 0 | 3
    Other substance use disorder | 0 | 0 | 0 | 0
Mental Health Mood Disorder Diagnosis [Count of Participants; unit: Participants] — Mental health mood disorder diagnoses (anxiety, depression) from the EHR
  Participants
    Anxiety | 46 | 35 | 46 | 127
    Depression | 40 | 42 | 37 | 119
General Anxiety Disorder Subscale of PHQ-4 (GAD 3+) [Count of Participants; unit: Participants] — General Anxiety Disorder (GAD) subscale of the Personalized Health Question (PHQ-4) in which higher values represent worst anxiety (range 0-6) and we categorize into having anxiety symptoms >=3 vs not having anxiety symptoms.
  Participants | 53 | 63 | 57 | 173
Personalized Health Questionnaire-2 (PHQ-2) (depression threshold of 3+) [Count of Participants; unit: Participants] — Personalized Health Question-2 (PHQ-2) in which higher values represent worst depression (range 0-6) and we categorize into having depression symptoms >=3 vs not having depression symptoms.
  Participants | 51 | 62 | 49 | 162
Roland Morris Disability Questionnaire-Revised [Mean (Standard Deviation); unit: units on a scale] — Roland Morris Disability Questionnaire Revised (RMDQ-R) assesses how low back pain affects functional activity. Higher scores indicate worst functional activity. Roland: Scale Range 0-24.
  units on a scale | 12.86 (5.5) | 13.49 (5.4) | 13.19 (5.5) | 13.18 (5.5)
Pain (PEG) [Mean (Standard Deviation); unit: units on a scale] — The PEG is a measure of pain (3-item composite score of P (pain intensity), E (pain interference with enjoyment in life), and G (pain interference with general activity). Higher scores indicate worse pain. PEG Scale Range: 0-10.
  units on a scale | 5.45 (2.2) | 6.06 (1.9) | 5.76 (2.0) | 5.85 (2.0)
Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Characteristic of Pain Intensity (single item in rating scale over last week 0-10)
  units on a scale | 5.73 (1.9) | 6.06 (1.9) | 5.76 (2.0) | 5.85 (2.0)
PROMIS Physical Function Subscale [Mean (Standard Deviation); unit: units on a scale] — Subscale that assesses physical function through a grading scale of activities of daily living. The PROMIS Physical Function scale is not a direct 0-100 scale; it uses a T-score scale with a population mean of 50 and a standard deviation of 10, where a higher score indicates better physical function.
  units on a scale | 38.31 (6.4) | 38.16 (6.5) | 38.14 (6.8) | 38.2 (6.6)
PROMIS Sleep Disturbance Subscale [Mean (Standard Deviation); unit: units on a scale] — Subscale that evaluates sleep quality and disturbances. The PROMIS Sleep Disturbance scale uses a T-score metric, not a 0-100 scale. A T-score of 50 represents the average sleep disturbance level for the U.S. general population, with a standard deviation of 10. A higher T-score indicates greater sleep disturbance.
  units on a scale | 53.1 (8.3) | 54.63 (8.6) | 53.14 (8.1) | 53.62 (8.3)
PROMIS Fatigue Subscale [Mean (Standard Deviation); unit: units on a scale] — Subscale that measures fatigue experience and impact. PROMIS Fatigue does not use a 0-100 scale for its T-score, but a T-score metric where 50 is the average for the U.S. general population. Scores above 50 indicate more fatigue than average.
  units on a scale | 55.19 (8.7) | 56.08 (9.0) | 54.75 (9.0) | 55.34 (8.9)
PROMIS Engagement in Social Roles Subscale [Mean (Standard Deviation); unit: units on a scale] — Measures ability to engage in social roles. A PROMIS T-score has a standardized mean of 50 and a standard deviation (SD) of 10. For measures related to social function, higher scores indicate better function and fewer limitations.
  units on a scale | 45.72 (8.2) | 45.14 (8.3) | 45.55 (8.5) | 45.48 (8.3)
Pain Catastrophizing [Mean (Standard Deviation); unit: units on a scale] — 13-item scale (0-52) in which higher scores indicate more pain catastrophizing.
  units on a scale | 9.12 (5.7) | 10.77 (5.9) | 9.45 (6.1) | 9.78 (5.9)
High Impact Chronic Pain [Count of Participants; unit: Participants] | 112 | 125 | 138 | 375
Sciatica [Count of Participants; unit: Participants] | 163 | 186 | 195 | 544
Expectations of Acupuncture [Mean (Standard Deviation); unit: units on a scale] — Measure of acupuncture expectation (1-10) in which higher scores indicate higher expectation.
  units on a scale | 6.36 (2.4) | 6.37 (2.4) | 6.38 (2.5) | 6.37 (2.4)
Sleep Duration [Mean (Standard Deviation); unit: hours] — Sleep duration (number of hours per night).
  hours | 6.52 (1.3) | 6.35 (1.5) | 6.44 (1.4) | 6.44 (1.4)
Fear Avoidance [Count of Participants; unit: Participants] — Fear avoidance of acupuncture.
  Participants | 49 | 50 | 51 | 150
Tobacco, Alcohol, Prescription Medication, and Other Substance User (TAPS) Tool [Count of Participants; unit: Participants]
  TAPS Positive Screen (Any Use) | 86 | 73 | 74 | 233
  Tobacco Use | 17 | 19 | 13 | 49
  Alcohol Use | 40 | 38 | 36 | 114
  Illicit Drug Use | 35 | 30 | 42 | 107
  Prescription Drug Use | 11 | 6 | 7 | 24
Self-Management Program [Count of Participants; unit: Participants] — Use of self-management program for back pain or other needs.
  Participants
    Back Pain | 23 | 21 | 30 | 74
    Other Needs | 8 | 4 | 3 | 15
    None | 234 | 240 | 235 | 709
Use of Mind-Body Techniques [Count of Participants; unit: Participants] — Use of mind-body techniques for back pain or other needs. Population: Missing data for 9 participants.
  Participants
    Back Pain: number analyzed (Participants) | 264 | 261 | 266 | 791
    Back Pain | 56 | 60 | 57 | 173
    Other Needs: number analyzed (Participants) | 264 | 261 | 266 | 791
    Other Needs | 29 | 25 | 31 | 85
    None: number analyzed (Participants) | 264 | 261 | 266 | 791
    None | 179 | 176 | 178 | 533
Use of Online Pain Management Program [Count of Participants; unit: Participants] — Use of online pain management program for back pain or other needs. Population: Missing data for 7 participants.
  Participants
    Back Pain: number analyzed (Participants) | 266 | 262 | 265 | 793
    Back Pain | 7 | 8 | 7 | 22
    Other Needs: number analyzed (Participants) | 266 | 262 | 265 | 793
    Other Needs | 3 | 0 | 0 | 3
    None: number analyzed (Participants) | 266 | 262 | 265 | 793
    None | 256 | 254 | 258 | 768
Psychological Counseling [Count of Participants; unit: Participants] — Use of psychological counseling for back pain or other needs. Population: Missing data for 4 participants
  Participants
    Back Pain: number analyzed (Participants) | 266 | 265 | 265 | 796
    Back Pain | 17 | 10 | 8 | 35
    Other Needs: number analyzed (Participants) | 266 | 265 | 265 | 796
    Other Needs | 4 | 3 | 4 | 11
    None: number analyzed (Participants) | 266 | 265 | 265 | 796
    None | 245 | 252 | 253 | 750
How has COVID affected your ability to get healthcare in the last 3 months? [Count of Participants; unit: Participants] — Population: Missing data for 5 participants
  Participants
    Reduced your ability to get healthcare a lot: number analyzed (Participants) | 265 | 263 | 267 | 795
    Reduced your ability to get healthcare a lot | 22 | 31 | 17 | 70
    Reduced your ability to get healthcare a little: number analyzed (Participants) | 265 | 263 | 267 | 795
    Reduced your ability to get healthcare a little | 59 | 47 | 61 | 167
    Not affected your ability to get healthcare: number analyzed (Participants) | 265 | 263 | 267 | 795
    Not affected your ability to get healthcare | 180 | 181 | 182 | 543
    Improved your ability to get healthcare: number analyzed (Participants) | 265 | 263 | 267 | 795
    Improved your ability to get healthcare | 4 | 4 | 7 | 15
How has COVID affected your overall health in the last 3 months? [Count of Participants; unit: Participants] — Population: Missing data for 9 participants
  Participants
    Your overall health is a lot worse: number analyzed (Participants) | 262 | 261 | 268 | 791
    Your overall health is a lot worse | 17 | 21 | 19 | 57
    Your overall health is a little worse: number analyzed (Participants) | 262 | 261 | 268 | 791
    Your overall health is a little worse | 81 | 85 | 72 | 238
    Not affected your overall health: number analyzed (Participants) | 262 | 261 | 268 | 791
    Not affected your overall health | 159 | 152 | 172 | 483
    Improved your overall health: number analyzed (Participants) | 262 | 261 | 268 | 791
    Improved your overall health | 5 | 3 | 5 | 13
Use of various types of pain relievers for Back Pain [Count of Participants; unit: Participants] — User of various types of pain relievers (NSAIDS, acetaminophen, cannabis, CBD only, herbal/nutritional supplements) for back pain.
  Participants
    NSAIDs | 161 | 155 | 171 | 487
    Acetaminophen | 148 | 174 | 162 | 484
    Cannabis | 50 | 53 | 59 | 162
    CBD Only | 47 | 48 | 42 | 137
    Herbal/Nutritional Supplements | 77 | 61 | 81 | 219
Weekly Exercise [Count of Participants; unit: Participants] — Exercise (active, low back, other movement) at least weekly.
  Participants
    Active Exercise | 179 | 190 | 195 | 564
    Low Back Exercise | 116 | 137 | 128 | 381
    Other Movement | 42 | 39 | 47 | 128
Weekly Exercise (number of days) [Mean (Standard Deviation); unit: Days] — Number of days of weekly exercise (active, low back, other movement).
  Days
    Weekly active exercise | 3.1 (2.7) | 3.24 (2.7) | 3.25 (2.6) | 3.2 (2.7)
    Weekly low back exercise | 2.02 (2.6) | 2.13 (2.6) | 2.19 (2.7) | 2.12 (2.7)
    Weekly other movement | .56 (1.6) | .42 (1.3) | .48 (1.4) | .49 (1.5)
3+ Days/Week of Exercise [Count of Participants; unit: Participants] — 3 or more days per week of exercise (active, low back, other movement).
  Participants
    3+ Days of Active Exercise | 145 | 146 | 157 | 448
    3+ Days of Low Back Exercise | 95 | 98 | 101 | 294
    3+ Days of Other Movement | 25 | 21 | 21 | 67
Roland Morris Disability Questionnaire Revised (RMDQ-R) - Back-Related Dysfunction (>=18 score) [Count of Participants; unit: Participants] — RMDQ-R assesses how low back pain affects functional activities. Higher scores indicate worst functional activity. Roland: Scale Range 0-24. This is a count of participants with back-related dysfunction score >=18 and participants with a score <18. This is a dichotomous variable to indicate high RDMQ scores. Scores generally indicate increasing severity, with 15-24 often considered moderate to severe, and scores above 18 (e.g., 19+) moving towards extreme disability or maximal impairment.
  Participants
    Roland Score >=18 | 59 | 70 | 67 | 196
    Roland Score <18 | 207 | 195 | 202 | 604

OUTCOME MEASURES:

1. Primary Outcome: Change in Back-related Disability at 6-month Post Randomization (Continuous)
Description: Change in back-related disability is defined as score change in Roland Morris Disability Questionnaire (RMDQ), a 24-item questionnaire which asked whether 24 specific activities were limited due to back pain during the past week. The RMDQ is scored from 0 to 24, with higher scores indicating more disability. Greater change between baseline and 6-months would indicate greater improvement.
Time Frame: Baseline to 6-month
Population: Participants were individuals >= 65 years of age with non-specific chronic low back pain (cLMP) persisting for >=3 months with pain-related interference (>= on general activity item from PEG) recruited from four different health systems. After baseline assessment, participants were randomized in equal proportions to the three arms. Participants completed follow-up assessments at 3-, 6-, and 12- months post-enrollment.
Measure: Least Squares Mean (95% Confidence Interval); unit: change in score from baseline on scale
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
change in score from baseline on scale | -2.1 [-2.7 to -1.5] | -3.1 [-3.7 to -2.5] | -3.6 [-4.3 to -3.0]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; Test type: Superiority; p = .024, Wald Test, 2-sided; Adjusted ANCOVA model for change from baseline fit with generalized estimating equations (GEE) with 3-, 6-, and 12-month in same model; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.9 to -0.1]
Statistical Analysis 2: Comparison: Usual Care vs Enhanced Acupuncture; Test type: Superiority; p = .001, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-2.5 to -0.6]
Statistical Analysis 3: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Test type: Superiority; p = .286, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.5 to 0.5]

2. Secondary Outcome: Change in Back-related Disability at 3-, and 12-month (Continuous)
Description: Change in back-related disability is defined as score change in RMDQ, a 24-item questionnaire which asked whether 24 specific activities were limited due to back pain during the past week. The RMDQ is scored from 0 to 24, with higher scores indicating more disability. Greater change between baseline and 3-months or 12-months would indicate greater improvement.
Time Frame: Test of Standard Acupuncture: Baseline to 3 months; Test of Maintenance effect: Baseline to 12 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score change from baseline on a scale
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
score change from baseline on a scale
  3 Months | -2.0 [-2.6 to -1.4] | -3.4 [-3.8 to -3.0] | -3.4 [-3.8 to -3.0]
  12 Months | -1.8 [-2.5 to -1.1] | -3.0 [-3.5 to -2.5] | -3.5 [-4.2 to -2.8]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 3 months; SA & EA are pooled because 3 months is considered standard acupuncture regardless of acupuncture treatment arm; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.1 to -0.7]
Statistical Analysis 2: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .008, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.1 to -0.3]
Statistical Analysis 3: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.6 to -0.7]
Statistical Analysis 4: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .27, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.4 to .4]

3. Secondary Outcome: Achieving Minimal Clinically Important Difference (MCID) in Back-related Disability at 3-, 6-, and 12-months (Binary)
Description: The MCID is measured by a 30% improvement (reduction) on the Roland Morris Disability Questionnaire Revised (RMDQ-R). The MCID reflects clinical improvement and estimates the percentage of individuals with a 30% improvement by intervention arm and 95% confidence intervals are adjusted means of a binary variables estimated using modified Poisson regression. Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702-6. doi: 10.1093/aje/kwh090. PMID: 15033648.
Time Frame: Study primary outcome timepoint: Baseline to 6 months; Test of Standard Acupuncture: Baseline to 3 months; Test of Maintenance effect: Baseline to 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: adjusted percentage of participants
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
adjusted percentage of participants
  3 Months | 29.9 [24.9 to 36.0] | 42.0 [38.0 to 46.4] | 42.0 [38.0 to 46.4]
  6 Months | 29.4 [24.3 to 35.5] | 39.1 [33.1 to 46.1] | 43.8 [38.0 to 50.4]
  12 Months | 28.4 [23.4 to 34.4] | 37.7 [33.6 to 42.3] | 43.8 [39.0 to 49.2]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < .001, Wald Test, 2-sided; Estimation performed with adjusted modified Poisson regression model with binary outcome, 30% improvement from baseline, fit with GEE; Risk Ratio (RR) = 1.40, 95% CI 2-sided [1.15 to 1.72]
Statistical Analysis 2: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .022, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.33, 95% CI 2-sided [1.04 to 1.70]
Statistical Analysis 3: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p < .001, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.49, 95% CI 2-sided [1.19 to 1.86]
Statistical Analysis 4: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .36, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.12, 95% CI 2-sided [.88 to 1.43]
Statistical Analysis 5: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .012, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.33, 95% CI 2-sided [1.06 to 1.66]
Statistical Analysis 6: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p < .001, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.54, 95% CI 2-sided [1.25 to 1.91]
Statistical Analysis 7: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .076, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.16, 95% CI 2-sided [.98 to 1.37]

4. Secondary Outcome: Change in Pain, Pain Interference With Enjoyment, General Activity (PEG) at 3-, 6- and 12-month (Continuous)
Description: Change in pain intensity and pain interference with enjoyment of life and general activity will be measured by PEG, a 3-item pain-intensity and pain-related interference composite measure assessing pain intensity, and pain interference with enjoyment of life and general activity. Each item is measured by a 0 to 10 scale with 10 indicating greater pain intensity or pain interference. The scores are then averaged with a higher average score indicating greater pain interference/intensity.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: change of score from baseline on a scale
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
change of score from baseline on a scale
  3 Months | -0.6 [-0.8 to -0.4] | -1.4 [-1.5 to -1.3] | -1.4 [-1.5 to -1.3]
  6 Months | -0.6 [-0.9 to -0.3] | -1.1 [-1.3 to -0.8] | -1.5 [-1.8 to -1.3]
  12 Months | -0.7 [-0.9 to -0.4] | -1.1 [-1.3 to -0.9] | -1.3 [-1.5 to -1.1]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.1 to -0.5]
Statistical Analysis 2: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .019, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.8 to -0.1]
Statistical Analysis 3: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.3 to -0.6]
Statistical Analysis 4: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .02, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.9 to -0.1]
Statistical Analysis 5: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .02, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.8 to -0.1]
Statistical Analysis 6: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1 to -0.3]
Statistical Analysis 7: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .22, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.6 to 0.1]

5. Secondary Outcome: Achieving MCID in Pain, Pain Interference With Enjoyment, General Activity (PEG) at 3-, 6-, and 12-months (Binary)
Description: The MCID is measured by a 30% improvement (reduction) on the PEG. The MCID reflects clinical improvement and estimates the percentage of individuals with a 30% improvement by intervention arm and 95% confidence intervals are adjusted means of a binary variables estimated using modified Poisson regression. Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702-6. doi: 10.1093/aje/kwh090. PMID: 15033648.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: adjusted percentage of participants
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
adjusted percentage of participants
  3 Months | 23.3 [18.7 to 29.1] | 41.1 [37.6 to 44.9] | 41.1 [37.6 to 44.9]
  6 Months | 29.4 [24.4 to 35.5] | 35.0 [30.5 to 40.2] | 40.5 [35.6 to 46.1]
  12 Months | 29.5 [24.5 to 35.5] | 35.9 [31.3 to 41.0] | 35.8 [30.4 to 42.2]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.76, 95% CI 2-sided [1.39 to 2.24]
Statistical Analysis 2: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .14, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.19, 95% CI 2-sided [.94 to 1.50]
Statistical Analysis 3: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .006, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.38, 95% CI 2-sided [1.10 to 1.73]
Statistical Analysis 4: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .167, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.16, 95% CI 2-sided [.94 to 1.42]
Statistical Analysis 5: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .089, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.22, 95% CI 2-sided [.97 to 1.52]
Statistical Analysis 6: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .12, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.21, 95% CI 2-sided [.95 to 1.55]
Statistical Analysis 7: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .99, Wald Test, 2-sided; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.00, 95% CI 2-sided [.80 to 1.25]

6. Secondary Outcome: Change in Physical Functioning at 3-, 6- and 12-month (Continuous)
Description: Change in the Patient-Reported Outcomes Measurement and Information System (PROMIS) Physical functioning short form 6b from the PROMIS-29 (6 items). The 6-item Physical function scale measures self-reported ability to perform activities rather than the actual performance of those activities. Each question has five response options, ranging from one to five. Raw scores range from 6 to 30, with higher scores indicating greater ability. The scores are then standardized using a T-score metric in which 50 is the reference mean and 10 is the standard deviation (SD) of that population.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: change in score from baseline on a scale
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
change in score from baseline on a scale
  3 Months | 0.8 [0.1 to 1.4] | 1.6 [1.2 to 2.1] | 1.6 [1.2 to 2.1]
  6 Months | 1.0 [0.4 to 1.7] | 1.2 [0.6 to 1.8] | 1.8 [1.2 to 2.5]
  12 Months | 1.0 [0.3 to 1.7] | 1.7 [1.0 to 2.3] | 1.5 [0.9 to 2.0]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .025, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .9, 95% CI 2-sided [.1 to 1.7]
Statistical Analysis 2: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .747, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .2, 95% CI 2-sided [-0.8 to 1.1]
Statistical Analysis 3: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .1, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .8, 95% CI 2-sided [-.1 to 1.7]
Statistical Analysis 4: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .22, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .6, 95% CI 2-sided [-.4 to 1.6]
Statistical Analysis 5: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .162, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .7, 95% CI 2-sided [-.3 to 1.6]
Statistical Analysis 6: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .277, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .5, 95% CI 2-sided [-.4 to 1.4]
Statistical Analysis 7: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .68, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.2, 95% CI 2-sided [-1 to .7]

7. Secondary Outcome: Patient Global Impression of Change (PGIC) at 3-, 6-, and 12- Months
Description: Patient Global Impression of Change in Overall Pain (1 item). This is a 0 to 6 scale ranging from much worse to much better, with higher scores indicating more improvement.
Time Frame: Study primary outcome timepoint: 6 months; Test of Standard Acupuncture: 3 months; Test of Maintenance effect: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in score from baseline on a scale
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
Change in score from baseline on a scale
  3 Months | 3.4 [3.2 to 3.5] | 4.5 [4.4 to 4.6] | 4.5 [4.4 to 4.6]
  6 Months | 3.3 [3.1 to 3.5] | 4.0 [3.8 to 4.1] | 4.6 [4.4 to 4.7]
  12 Months | 3.3 [3.1 to 3.6] | 3.9 [3.7 to 4.1] | 4.1 [4.0 to 4.3]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.9 to 1.4]
Statistical Analysis 2: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .7, 95% CI 2-sided [.4 to 1]
Statistical Analysis 3: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [1 to 1.5]
Statistical Analysis 4: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .6, 95% CI 2-sided [.3 to .9]
Statistical Analysis 5: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .5, 95% CI 2-sided [.2 to .8]
Statistical Analysis 6: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .8, 95% CI 2-sided [.5 to 1.1]
Statistical Analysis 7: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .06, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .3, 95% CI 2-sided [0 to 0.5]

8. Secondary Outcome: Serious Adverse Effects (SAE)/Non-Serious Adverse Effects (AE)
Description: Serious adverse events were defined as hospitalizations and deaths. Only potentially treatment-related non-serious adverse events were reported in the acupuncture arms (not usual care).
Time Frame: SAE: 12 months from electronic health record data; AE: 12 months from acupuncture treatment records and follow-up interviews.
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
events
  Serious Adverse Events (SAEs) | 18 | 24 | 24
  Adverse Events (AEs) | 0 | 24 | 27

9. Other Pre Specified Outcome: Change in Sleep Quality
Description: Change in sleep quality is measured by the six-item Patient-Reported Outcomes Measurement and Information System (PROMIS) Sleep Disturbance Short Form 6a. The raw computed score has a range of 6-30 with higher scores indicating more sleep disturbance. The raw score is converted to a T-score with mean of 50, standard deviation of 10. Higher T-scores indicate worse sleep quality. PROMIS Sleep Scoring Manual. Published online June 3, 2022. https://www.healthmeasures.net/images/PROMIS/manuals/Scoring_Manual_Only/PROMIS_Sleep_Scoring_Manual_03June2022.pdf
Time Frame: Study primary outcome timepoint: Baseline to 6 months (sleep quality)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in T-score from baseline
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
Change in T-score from baseline | -1.18 [-2.14 to -0.22] | -1.62 [-2.4 to -0.84] | -2.19 [-3.17 to -1.22]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = -.06, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.7 to .08]
Statistical Analysis 2: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = -.15, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1, 95% CI 2-sided [-2.4 to .3]
Statistical Analysis 3: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .387, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.6, 95% CI 2-sided [-1.9 to .7]

10. Other Pre Specified Outcome: Change in Sleep Duration at 3-, 6- and 12-month
Description: Change in 1-item sleep duration scale for sleep duration.
Time Frame: Study primary outcome timepoint: Baseline to 6 months (sleep duration); Test of Standard Acupuncture: Baseline to 3 months (sleep duration only); Test of Maintenance effect: Baseline to 12 months (sleep duration only)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: change in hours from baseline
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
change in hours from baseline
  3 Months | 0.17 [0.03 to 0.31] | 0.17 [0.08 to 0.26] | 0.17 [0.08 to 0.26]
  6 Months | 0.02 [-0.1 to 0.15] | 0.12 [0.0 to 0.25] | 0.2 [0.08 to 0.32]
  12 Months | 0.13 [-0.1 to 0.27] | 0.18 [0.04 to 0.31] | 0.27 [0.16 to 0.37]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .967, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0, 95% CI 2-sided [-.02 to .02]
Statistical Analysis 2: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .272, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .1, 95% CI 2-sided [-.1 to .3]
Statistical Analysis 3: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .049, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .2, 95% CI 2-sided [0 to 0.4]
Statistical Analysis 4: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .409, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .1, 95% CI 2-sided [-.1 to .3]
Statistical Analysis 5: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .62, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0, 95% CI 2-sided [-.1 to .2]
Statistical Analysis 6: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .121, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .1, 95% CI 2-sided [0 to .3]
Statistical Analysis 7: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .27, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .1, 95% CI 2-sided [-.1 to .2]

11. Other Pre Specified Outcome: Change in Symptoms Suggesting Clinically Relevant Anxiety at 3-, 6- and 12-month (Continuous)
Description: Change in PRO scores about the frequency of being anxious or having uncontrollable worry over the past two weeks from the GAD-2, which is part of the PHQ-4. Each item is measured by a 0 to 3 scale with 3 indicating greater anxiety. GAD-2 range is 0-6, with 6 being greater anxiety symptoms.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: change in score from baseline on a scale
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
change in score from baseline on a scale
  3 Months | 0.0 [-0.1 to 0.2] | -0.2 [-0.3 to 0.0] | -0.2 [-0.3 to 0.0]
  6 Months | 0.1 [-0.2 to 0.3] | -0.3 [-0.4 to -0.1] | -0.2 [-0.4 to 0.0]
  12 Months | 0.0 [-0.2 to 0.2] | -0.4 [-0.5 to -0.3] | -0.3 [-0.4 to -0.1]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .069, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.2, 95% CI 2-sided [-.4 to .02]
Statistical Analysis 2: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .013, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.3, 95% CI 2-sided [-.6 to -.1]
Statistical Analysis 3: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .043, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.3, 95% CI 2-sided [-.5 to -.1]
Statistical Analysis 4: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .629, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .1, 95% CI 2-sided [-.2 to .3]
Statistical Analysis 5: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .001, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.4, 95% CI 2-sided [-.6 to -.2]
Statistical Analysis 6: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .019, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.3, 95% CI 2-sided [-.5 to -.05]
Statistical Analysis 7: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .271, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .1, 95% CI 2-sided [-.1 to .3]

12. Other Pre Specified Outcome: Change in Symptoms Suggesting Depression at 3-, 6- and 12-month (Continuous)
Description: Change in PRO scores about the frequency of depressed mood and anhedonia over the past two weeks from the PHQ-2. Each item is measured by a 0 to 3 scale with 3 indicating greater depression. Total score is 0-6, with 6 indicating greater depression.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: change in score from baseline on a scale
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
change in score from baseline on a scale
  3 Months | 0.0 [-0.2 to 0.1] | -0.2 [-0.3 to -0.1] | -0.2 [-0.3 to -0.1]
  6 Months | 0.0 [-0.2 to 0.2] | -0.2 [-0.4 to -0.1] | -0.3 [-0.4 to -0.1]
  12 Months | -0.2 [-0.4 to -0.1] | -0.4 [-0.5 to -0.3] | -0.3 [-0.4 to -0.2]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .191, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.1, 95% CI 2-sided [-.3 to .1]
Statistical Analysis 2: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .038, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.3, 95% CI 2-sided [-.5 to -.01]
Statistical Analysis 3: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .019, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.3, 95% CI 2-sided [-.5 to -.05]
Statistical Analysis 4: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .803, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.03, 95% CI 2-sided [-.2 to .2]
Statistical Analysis 5: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .163, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.2, 95% CI 2-sided [-.4 to .1]
Statistical Analysis 6: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .625, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.05, 95% CI 2-sided [-.2 to .1]
Statistical Analysis 7: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .198, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .1, 95% CI 2-sided [-.1 to .3]

13. Other Pre Specified Outcome: Change in Fatigue at 3-, 6- and 12-month (Continuous)
Description: Change in fatigue will be measured by a change in T-score of the 4-item Patient-Reported Outcomes Measurement and Information System (PROMIS) Fatigue Subscale - SF 4a. This PROMIS measure has a T-score with a mean of 50 and a standard deviation of 10, meaning a score of 50 is average. Higher T-scores indicates greater fatigue. PROMIS Fatigue Scoring Manual. Published online November 4, 2016. https://www.fda.gov/media/137977/download
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: change in T-score from baseline
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
change in T-score from baseline
  3 Months | -2.42 [-3.43 to -1.41] | -3.27 [-4.09 to -2.46] | -3.27 [-4.09 to -2.46]
  6 Months | -1.55 [-2.61 to -0.48] | -2.06 [-3.14 to -0.97] | -2.52 [-3.69 to -1.35]
  12 Months | -1.18 [-2.24 to -0.12] | -2.47 [-3.39 to -1.54] | -3.50 [-4.26 to -2.74]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .194, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.9, 95% CI 2-sided [-2.1 to .4]
Statistical Analysis 2: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .51, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.5, 95% CI 2-sided [-2 to 1]
Statistical Analysis 3: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .218, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1, 95% CI 2-sided [-2.5 to .6]
Statistical Analysis 4: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .62, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.5, 95% CI 2-sided [-2.3 to 1.4]
Statistical Analysis 5: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .07, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.7 to .1]
Statistical Analysis 6: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = 0, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-3.6 to -1]
Statistical Analysis 7: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .086, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1, 95% CI 2-sided [-2.2 to .1]

14. Other Pre Specified Outcome: Change in Ability to Engage in Social Roles at 3-, 6- and 12-month (Continuous)
Description: Change in ability to engage in social roles will be measured by the 4-item subscale for ability to participate in social roles in PROMIS. PROMIS measures are standard T-score range of 20-80, with higher scores indicating greater ability to engage in social roles.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: change in score from baseline on a scale
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
Number analyzed (Participants) | 266 | 265 | 269
change in score from baseline on a scale
  3 Months | 0.4 [-0.5 to 1.2] | 1.6 [1.0 to 2.2] | 1.6 [1.0 to 2.2]
  6 Months | 0.5 [-0.4 to 1.4] | 1.3 [0.5 to 2.1] | 1.6 [0.5 to 2.6]
  12 Months | -0.2 [-1.0 to 0.6] | 1.6 [0.9 to 2.3] | 1.4 [0.6 to 2.1]
Statistical Analysis 1: Comparison: Usual Care vs Standard Acupuncture; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .023, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [.2 to 2.3]
Statistical Analysis 2: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .186, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .8, 95% CI 2-sided [-.4 to 2]
Statistical Analysis 3: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .107, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-.2 to 2.5]
Statistical Analysis 4: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 6 months; Test type: Superiority; p = .651, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .3, 95% CI 2-sided [-1 to 1.7]
Statistical Analysis 5: Comparison: Usual Care vs Standard Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .001, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [.7 to 2.9]
Statistical Analysis 6: Comparison: Usual Care vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .007, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [.4 to 2.7]
Statistical Analysis 7: Comparison: Standard Acupuncture vs Enhanced Acupuncture; Difference in change from baseline at 12 months; Test type: Superiority; p = .656, Wald Test, 2-sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.2, 95% CI 2-sided [-1.2 to .8]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the one-year period of enrollment for each study participant.
Description: Adverse events were identified by acupuncturists, follow-up mailers and ad-hoc participant reports.
  Serious adverse events, defined as hospitalizations and deaths, were assessed monthly from the electronic health record (EHR) and medical-record abstraction conduction by physician monitors at each site to determine relatedness.
  We collected only potentially treatment-related non-serious adverse events in the acupuncture arms (not in usual care).
Arm/Group | Usual Care | Standard Acupuncture | Enhanced Acupuncture
All-Cause Mortality (participants affected / at risk) | 2/266 | 0/265 | 1/269
Serious Adverse Events (participants affected / at risk) | 18/266 | 24/265 | 24/269
Other Adverse Events (participants affected / at risk) | 0/266 | 24/265 | 27/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=266) | Standard Acupuncture (N=265) | Enhanced Acupuncture (N=269)
Acute Encephalopathy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Anemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Arrythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bladder Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bradycardia and syncope (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Car Accident (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Collapsed Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
COVID (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
COVID (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Death (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Difficulty passing food (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysautonomia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis and Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Heart Attack (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hip Fracture (General disorders) | 0 (0) | 2 (2) | 0 (0)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal Infection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Medication Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Myasthenia Gravis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Pinched Nerve (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Rib and cervical spine fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) — Includes sepsis, septic arthritis, and septic shock
Small bowel obstruction (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Stomach ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Vascular disorders) | 3 (4) | 3 (3) | 1 (1)
Surgical procedure (Surgical and medical procedures) | 2 (2) | 5 (5) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=266) | Standard Acupuncture (N=265) | Enhanced Acupuncture (N=269)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Low Back Pain (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) | 0 (0)
Lower Extremity Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 4 (5)
Pain at Needle Insertion Site (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 11 (14)
Swelling at Needle Insertion Site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Broken Ribs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bruising at Needle Injection Site (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Falling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Generalized Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
High Blood Pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Low Back Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lower Extremity Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lower Extremity Numbness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lower Extremity Pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Muscle Spasm at Needle Insertion Site (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Neck Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Nerve Pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nerve Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Periorbital Swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postural Instability (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Spinal Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Warmth at Needle Insertion Site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations: UMC control group precludes assessment of attention or other nonspecific effects on outcomes; results may be affected by subjectivity in PROs; treatment impact on medication changes unattainable due to limited robust medication-dispensing data at 2 sites; even after imputation and non-response weighting, residual bias may remain, potentially due to differential loss to follow-up by arm; significant findings for secondary outcomes should be interpreted cautiously.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT04982315/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT04982315/SAP_001.pdf